CLINICAL TRIAL: NCT06757972
Title: Effect of Tele Rehabilitation in Breaking Barriers With Mobility Impairments in Rural Areas: a Randomized Controlled Trial
Brief Title: Effect of Tele Rehabilitation in Breaking Barriers With Mobility Impairments in Rural Areas (RCT)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/751
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Mobility Limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group I (Experimental)
  Interventions: Combination Product: Tele Rehab
- Interventional group II (Active Comparator)
  Interventions: Diagnostic Test: Formal Rehab

INTERVENTIONS:
Combination Product: Tele Rehab — Tele rehabilitation intervention is 6 months standardized program aimed to provide special rehabilitation services to patients with mobility impairments in rural areas without the need for them to travel to healthcare facility in big cities. The program consists of standard exercises addressing key components of mobility impairments.
  Arms: Interventional group I
Diagnostic Test: Formal Rehab — After formal rehabilitation is completed, some impaired mobility victims re-access services; no attempt will be made to stop the control group from accessing further care, in either a public or private setting. However, physical activity participation will be assured during monthly phone call by a blinded -research assistant. Participants in this group will undergo three assessments at baseline, 6 and 12 months
  Arms: Interventional group II

SUMMARY:
Tele-rehabilitation offers remote healthcare services via telecommunication technology to patients who face challenges in accessing traditional in-person rehabilitation. This randomized controlled trial investigated the effectiveness of tele-rehabilitation in overcoming mobility impairments in rural Pakistan.

DETAILED DESCRIPTION:
A total of 92 participants, equally divided into intervention and control groups, were assessed. The intervention group received a 6-month tele-rehabilitation program, including video consultations, home visits, structured calls, and text messages.

ELIGIBILITY:
Inclusion Criteria:

* People will be eligible for participation if they have had any disorder causing mobility impairment,
* Lives in rural areas,
* Are over the age of 20,
* Have been discharged from inpatient, outpatient and community physiotherapy living in their home, (Saywell, Vandal et al. 2012)
* Have medical approval from their general practitioner to engage in low to medium level exercise programs,
* At least 3 score on telephone cognitive screening questionnaire (Callahan, Unverzagt et al. 2002)
* Have limitation in mobility, physical function of arm, leg or both.

Exclusion Criteria:

* If they have confirmed cerebellar or brain stem stroke,
* Tele rehabilitation involvement require frequent communication with physiotherapist so using interpreter is considered impractical,
* Participants enrolled in other rehabilitation programs,
* Lack of necessary devices (e.g, internet, smartphone, tablet, computer) for tele rehabilitation.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | 12 Months
  The scale consists of 14 tasks that a healthcare provider scores on a scale from 0 to 4. The higher the score, the better your balance. It's a straightforward, reliable test providers use to assess functional balance
Quality of Life (QOL) | 12 Months
  The QOLS scores are summed so that a higher score indicates higher quality of life. Average total score for healthy populations is about 90.

CONTACTS AND LOCATIONS:
Locations (1):
- Superior University CRC, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No